CLINICAL TRIAL: NCT01798602
Title: Collaborative H1N1 Adjuvant Treatment (CHAT) Pilot Trial
Acronym: CHAT Pilot
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: H1N1 pandemic concluded
Sponsor: Canadian Critical Care Trials Group (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCCTG
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: H1N1 Influenza
Keywords: H1N1; Rosuvastatin
MeSH Terms: conditions — Orthomyxoviridae Infections | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 40 mg via nasogastric tube then 20 mg po or via nasogastric tube daily for 14 days or until hospital discharge Placebo is identical capsule with no active drug
  Both are crushed for administration
  Interventions: Drug: Rosuvastatin or identical placebo
- Placebo (Placebo Comparator): Identical drug vehicle with no active agent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin or identical placebo — Tablet crushed for administration via feeding tube
  Other Names: Crestor; Placebo
  Arms: Rosuvastatin
Drug: Placebo — Identical placebo for rosuvastatin
  Arms: Placebo

SUMMARY:
The CHAT Pilot Trial is designed to compare rosuvastatin against placebo in patients with suspected H1N1. The pilot study will assess the feasibility of our clinical protocols, and study procedures.

DETAILED DESCRIPTION:
This trial is a pilot study to assess the feasibility and acceptability of a double blind randomized controlled trial (RCT) evaluating the efficacy of rosuvastatin as adjuvant therapy for H1N1 influenza

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adult patients > 16 years of age admitted to an adult ICU for any reason with suspected, probable or confirmed novel swine origin influenza A/H1N1 infection
* Requiring mechanical ventilation (invasive or non-invasive)
* Receiving antiviral therapy (any medication at any dose and for any intended duration) for < 72 hours
* Clinicians must have a 'moderate', 'high' or 'moderate to high' index of suspicion for H1N1

Exclusion Criteria:

* Age < 16 years
* Do not resuscitate or re-intubate order documented on chart or anticipated withdrawal of life support
* Weight < 40 kg
* Unable to receive or unlikely to absorb enteral study drug (e.g. incomplete or complete bowel obstruction, intestinal ischemia, infarction, short bowel syndrome)
* Rosuvastatin specific exclusions:

  1. Already receiving a statin (Atorvastatin, Lovastatin, Simvastatin, Pravastatin, Rosuvastatin)
  2. Allergy or intolerance to statins
  3. Receiving niacin, fenofibrate, cyclosporine, gemfibrozil, lopinavir, ritonavir or planned use of oral contraceptives or estrogen therapy during the ICU stay
  4. CK exceeds 10 times ULN or ALT exceeds 8 times the ULN
* Severe chronic liver disease (Child-Pugh Score 11-15) (see Appendix 6)
* Previous enrolment in this trial
* Pregnancy or breast feeding
* At the time of enrolment, patients must not have received >72 hours of antiviral therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible patients enrolled in the CHAT study | Over 6 month period or during H1N1 pandemic
  This was a pilot study whose primary goal was to evaluate the feasibility of patient recruitment during an emerging pandemic

SECONDARY OUTCOMES:
Adherence to the medication administration regimen as outlined in the study protocol. | 2 weeks
Proportion of completed primary and secondary endpoints for the planned full CHAT trial that are collected. | 6 months
The number of study withdrawals due to administration of open label statins and withdrawals of consent. | Up to 28 days or until hospital discharge
Recruitment rates by consent model. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Burns KE, Chant C, Smith O, Cuthbertson B, Fowler R, Cook DJ, Kruger P, Webb S, Alhashemi J, Dominguez-Cherit G, Zala C, Rubenfeld GD, Marshall JC. A Canadian Critical Care Trials Group project in collaboration with the international forum for acute care trialists - Collaborative H1N1 Adjuvant Treatment pilot trial (CHAT): study protocol and design of a randomized controlled trial. Trials. 2011 Mar 9;12:70. doi: 10.1186/1745-6215-12-70. PMID 21388549
- See also: International Forum for Acute Care Trialists Website — http://www.infactglobal.org
- See also: Canadian Critical Care Trials Group — http://www.ccctg.ca